CLINICAL TRIAL: NCT04526509
Title: Master Protocol to Assess the Safety and Recommended Phase 2 Dose of Next Generations of Autologous Enhanced NY-ESO-1/ LAGE-1a TCR Engineered T-cells, Alone or in Combination With Other Agents, in Participants With Advanced Tumors
Brief Title: Master Protocol to Assess Safety and Dose of First Time in Human Next Generation Engineered T Cells in NY-ESO-1 and/or LAGE-1a Positive Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a change in GSK's R&D priorities.
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209012; 2019-004446-14 (EudraCT Number)
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms
Keywords: Adoptive T-cell therapy; Advanced synovial sarcoma; Advanced non-small cell lung cancer; Advanced tumors; GSK3845097; GSK3901961; GSK4427296; T cell receptors; Leukapheresis; Advanced myxoid/round cell liposarcoma
MeSH Terms: conditions — Neoplasms; Liposarcoma, Myxoid | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Masking Description: This will be an open-label study. Hence, there will be no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Substudy 1: Cohort 1 - GSK3901961 in previously treated metastatic NSCLC (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive GSK3901961, as intravenous (IV) infusion after completing lymphodepleting chemotherapy.
  Interventions: Drug: GSK3901961; Drug: Cyclophosphamide; Drug: Fludarabine
- Substudy 1: Cohort 2 - GSK3901961 in previously treated advanced SS or MRCLS (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive GSK3901961, as IV infusion after completing lymphodepleting chemotherapy.
  Interventions: Drug: GSK3901961; Drug: Cyclophosphamide; Drug: Fludarabine
- Substudy 2: GSK3845097 in previously treated advanced SS or MRCLS (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive GSK3845097, as IV infusion after completing lymphodepleting chemotherapy.
  Interventions: Drug: GSK3845097; Drug: Cyclophosphamide; Drug: Fludarabine
- Substudy 3: GSK4427296 in previously treated advanced SS or MRCLS (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive GSK4427296, as IV infusion after completing lymphodepleting chemotherapy.
  Interventions: Drug: GSK4427296; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: GSK3901961 — GSK3901961 as an IV infusion.
  Arms: Substudy 1: Cohort 1 - GSK3901961 in previously treated metastatic NSCLC; Substudy 1: Cohort 2 - GSK3901961 in previously treated advanced SS or MRCLS
Drug: GSK3845097 — GSK3845097 as an IV infusion.
  Arms: Substudy 2: GSK3845097 in previously treated advanced SS or MRCLS
Drug: GSK4427296 — GSK4427296 as an IV infusion.
  Arms: Substudy 3: GSK4427296 in previously treated advanced SS or MRCLS
Drug: Cyclophosphamide — Cyclophosphamide will be used as lymphodepleting chemotherapy and will be administered via IV route.
Drug: Fludarabine — Fludarabine will be used as lymphodepleting chemotherapy and will be administered via IV route.

SUMMARY:
This trial will evaluate the safety and efficacy of first time in human engineered T-cell therapies, in participants with advanced tumors.

DETAILED DESCRIPTION:
This study is a master protocol. It has two sub studies registered as 209012 Sub Study 1 (NCT06048705) and 209012 Sub Study 2 (NCT05943990).

ELIGIBILITY:
Eligibility Criteria:

Inclusion criteria:

* Participant must be >=18 years of age and weighs ≥40 kg on the day of signing informed consent
* Participant must be positive for HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 alleles
* Participant's tumor must have tested positive for NY-ESO-1 and/or LAGE-1a expression by a GSK designated laboratory
* Performance status: Eastern Cooperative Oncology Group of 0-1
* Participant must have adequate organ function and blood cell counts 7 days prior to leukapheresis
* Participant must have measurable disease according to RECIST v1.1.

Additional criteria for participants with SS/ MRCLS:

* Participant has advanced (metastatic or unresectable) SS or MRCLS confirmed by local histopathology with evidence of disease-specific translocation
* Participant has completed at least one standard of care (SOC) treatment including anthracycline containing regimen unless intolerant to or ineligible to receive the therapy. Participants who are not candidates to receive anthracycline should have received ifosfamide unless also intolerant to or ineligible to receive ifosfamide. Participants who received neoadjuvant/adjuvant anthracycline or ifosfamide based therapy and progressed will be eligible

Additional criteria for participants with non-small cell lung cancer (NSCLC):

* Participant has Stage IV NSCLC as confirmed by histology or cytology
* Prior therapies for participants lacking actionable genetic aberrations (i.e., wild type), per National Comprehensive Cancer Network (NCCN) guidelines: participant has been previously treated with or is intolerant to programmed death receptor-1 (PD)-1/Programmed death ligand 1 (PD-L1) checkpoint blockade therapy and has been previously treated with or is intolerant to a platinum-based chemotherapy. Adjuvant therapy will count as a regimen if completed within 6 months before relapse. Or for participants that harbors an actionable genetic aberration (e.g. BRAF, anaplastic lymphoma kinase [ALK]/ c-ros oncogene 1 [ROS1] etc.), per NCCN guidelines: participants has been previously treated with or is intolerant to SOC therapy, including targeted therapy, as recommended by NCCN or equivalent country-level guidelines (European Society for Medical Oncology [ESMO], National Institute for Health & Care Excellence [NICE]) . Or Investigator has decided that additional lines of SOC therapy after the first line are not in the participant's best interest.

Exclusion criteria:

* Central nervous system (CNS) metastases, with certain exceptions for CNS metastases in NSCLC as specified in the protocol
* Any other prior malignancy that is not in complete remission
* Clinically significant systemic illness
* Prior or active demyelinating disease
* History of chronic or recurrent (within the last year prior to leukapheresis) severe autoimmune or immune mediated disease requiring steroids or other immunosuppressive treatments
* Previous treatment with genetically engineered NY-ESO-1-specific T cells, NY-ESO-1 vaccine or NY-ESO-1 targeting antibody
* Prior gene therapy using an integrating vector
* Previous allogeneic hematopoietic stem cell transplant within the last 5 years or solid organ transplant
* Washout periods for prior radiotherapy and systemic chemotherapy must be followed
* Major surgery within 4 weeks prior to lymphodepletion
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adaptimmune Patient Enquiries, Principal Investigator — Adaptimmune
Locations (16):
- United States (8):
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Melbourne, Victoria, Australia
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Germany (3):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
- GSK Investigational Site, Amsterdam, Netherlands
- GSK Investigational Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This master protocol study includes results data of screened participants for all the sub studies (NCT06048705 and NCT05943990). Results data is presented separately for 209012 Sub Study 1 (NCT06048705) and 209012 Sub Study 2 (NCT05943990). No participants were recruited for Sub Study 3. This is a master record and only contains data during screening phase (Day -35 to Day -8)
Pre-assignment Details: This study and the sub studies associated were terminated due to a change in GSK's R&D priorities.
Groups:
- All Screened Participants: Participants with advanced tumors were screened for HLA/NY-ESO-1 expression
- Sub Study 1 (NCT06048705)-GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells: Eligible participants were leukapheresed to manufacture engineered T cells. Participants then received 1 × 10^9 - 8 × 10^9 cells of GSK3901961 as an intravenous (IV) infusion in two aliquots (approximately 30% on Day 1 and approximately 70% on Day 8) for sentinel participant after completing lymphodepleting chemotherapy regimen that generally consisted of 30 milligram (mg)/meter (m)^2/day fludarabine for 4 days (Day -7 to -4) and 900mg/ m^2/day cyclophosphamide for 3 days (Day -6 to -4).
- Sub Study 1 (NCT06048705) GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells: Eligible participants were leukapheresed to manufacture engineered T cells. Participants then received 0.1 × 10^9 - 0.8 × 10^9 cells of GSK3901961 as an intravenous (IV) infusion on Day 1 after completing lymphodepleting chemotherapy regimen that generally consisted of 30 milligram (mg)/meter (m)^2/day fludarabine for 4 days (Day -7 to -4) and 900mg/ m^2/day cyclophosphamide for 3 days (Day -6 to -4).
- Sub Study 1 (NCT06048705)-No Treatment: No Treatment arm consisted of participants who underwent leukapheresis but did not go on to receive lymphodepletion chemotherapy and T cell infusion.
- Sub Study 2 (NCT05943990)-GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells: Eligible participants were leukapheresed to manufacture engineered T cells. Participants then received 1 × 10^9 - 8 × 10^9 cells of GSK3845097 as an intravenous (IV) infusion in two aliquots (approximately 30% on Day 1 and approximately 70% on Day 8) for sentinel participants or all at once on Day 1 for all other participants after completing lymphodepleting chemotherapy regimen that generally consisted of 30 milligram (mg)/meter (m)^2/day fludarabine for 4 days (Day -7 to -4) and 900mg/ m^2/day cyclophosphamide for 3 days (Day -6 to -4).
- Sub Study 2 (NCT05943990)-GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells: Eligible participants were leukapheresed to manufacture engineered T cells. Participants then received 0.1 × 10^9 - 0.8 × 10^9 cells of GSK3845097 as an intravenous (IV) infusion on Day 1 after completing lymphodepleting chemotherapy regimen that generally consisted of 30 milligram (mg)/meter (m)^2/day fludarabine for 4 days (Day -7 to -4) and 900mg/ m^2/day cyclophosphamide for 3 days (Day -6 to -4).
- Sub Study 2 (NCT05943990)-No Treatment: No Treatment arm consists of participants who underwent leukapheresis but did not go on to receive lymphodepletion chemotherapy and T cell infusion.
Period: Screening (Day -35 to Day -8)
Arm/Group | All Screened Participants | Sub Study 1 (NCT06048705)-GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | Sub Study 1 (NCT06048705) GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | Sub Study 1 (NCT06048705)-No Treatment | Sub Study 2 (NCT05943990)-GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | Sub Study 2 (NCT05943990)-GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | Sub Study 2 (NCT05943990)-No Treatment
Started (Participants consented to HLA/NY-ESO-1 target expression screening) | 327 | 0 | 0 | 0 | 0 | 0 | 0
Participants Were Tested for HLA-type | 277 (277 participants were tested for HLA-type) | 0 | 0 | 0 | 0 | 0 | 0
Participants Tested for HLA-type and Were HLA Positive | 146 (146 participants were HLA positive for A*02:01, A*02:05 or A*02:06 alleles) | 0 | 0 | 0 | 0 | 0 | 0
Participants Tested HLA Positive and NY-ESO-1 Expression Positive | 49 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Participants deemed eligible and enrolled) | 12 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 315 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not tested for both HLA-type and NY-ESO-1 tumor expression | 40 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Tested for NY-ESO-1 tumor expression but not HLA-type and were NY-ESO-1 negative | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Tested for NY-ESO-1 but not HLA-type and were NY-ESO-1 positive but not met other inclusion criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Tested for HLA-type and were HLA negative | 131 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Tested HLA positive and were NY-ESO-1 Negative or Not Evaluable | 97 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — HLA and NY-ESO-1 expression positive but not enrol in the study due to study terminated by sponsor | 23 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — HLA and NY-ESO-1 expression positive and did not meet inclusion/exclusion criteria | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — HLA and NY-ESO-1 expression positive and did not enrol due to physician decision | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — HLA and NY-ESO-1 expression positive and did not enrol as met eligibility criteria but not needed | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — HLA and NY-ESO-1 expression positive and did not enrol due to withdrawal by participant | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Enrolled
Arm/Group | All Screened Participants | Sub Study 1 (NCT06048705)-GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | Sub Study 1 (NCT06048705) GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | Sub Study 1 (NCT06048705)-No Treatment | Sub Study 2 (NCT05943990)-GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | Sub Study 2 (NCT05943990)-GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | Sub Study 2 (NCT05943990)-No Treatment
Started | 0 (12 participants who completed screening period were enrolled to Sub Studies 1 and 2) | 1 | 4 | 2 | 2 | 2 | 1
Completed (Participants who received T cell infusion and were followed up in this study until death or until transfer to the separate long term follow-up study are considered to have completed.) | 0 | 0 | 4 (2 participants died and 2 participants were transferred to the separate long term follow-up study 208750 (NCT03391778).) | 0 | 2 (2 participants were transferred to separate long term follow-up study 208750 (NCT03391778)) | 2 (2 participants died.) | 0
Not Completed | 0 | 1 | 0 | 2 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death prior to lymphodepletion | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Did not meet Inclusion/Exclusion Criteria | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population that included all participants who started leukapheresis procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sub Study 1 (NCT06048705)-GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | Sub Study 1 (NCT06048705) GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | Sub Study 1 (NCT06048705)-No Treatment | Sub Study 2 (NCT05943990)-GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | Sub Study 2 (NCT05943990)-GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | Sub Study 2 (NCT05943990)-No Treatment | Total
Number analyzed (Participants) | 1 | 4 | 2 | 2 | 2 | 1 | 12
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  19-64 years | 1 | 3 | 2 | 2 | 1 | 1 | 10
  >=65 years | 0 | 1 | 0 | 0 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 0 | 0 | 3
  Male | 0 | 3 | 1 | 2 | 2 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 4 | 2 | 2 | 2 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 1 | 4 | 2 | 1 | 2 | 1 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 2 | 1 | 0 | 1 | 1 | 5
  Sweden | 0 | 1 | 0 | 0 | 1 | 0 | 2
  United States | 1 | 0 | 1 | 2 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled Across Sub Studies
Description: Number of Participants Randomized across sub studies are presented.
Time Frame: Day -7
Population: Screened Population includes all participants who signed an ICF to participate in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Screened Participants
Number analyzed (Participants) | 327
Participants
  Sub Study 1 | 7
  Sub Study 2 | 5

ADVERSE EVENTS:
Time Frame: Screening (Day -35 to Day -8)
Description: Adverse events were not collected during screening.
Arm/Group | All Screened Participants | Sub Study 1 (NCT06048705)-GSK3901961 1 × 10^9 - 8 × 10^9 Transduced Cells | Sub Study 1 (NCT06048705) GSK3901961 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | Sub Study 1 (NCT06048705)-No Treatment | Sub Study 2 (NCT05943990)-GSK3845097 1 × 10^9 - 8 × 10^9 Transduced Cells | Sub Study 2 (NCT05943990)-GSK3845097 0.1 × 10^9 - 0.8 × 10^9 Transduced Cells | Sub Study 2 (NCT05943990)-No Treatment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT04526509/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT04526509/SAP_001.pdf